CLINICAL TRIAL: NCT07336199
Title: Pairing Subjective Patient Rating and Local Field Potentials for DBS Programming
Brief Title: Pairing Subjective Patient Rating and DBS Programming
Acronym: PERCEPT-DBS
Status: Recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Thomas Köglsperger, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: PERCEPT-DBS STUDY
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease (PD)
MeSH Terms: conditions — Parkinson Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Parkinson's disease patients with STN-DBS (PERCEPT-DBS cohort): Patients with idiopathic Parkinson's disease who have undergone bilateral deep brain stimulation (DBS) of the subthalamic nucleus (STN). Participants are implanted with sensing-enabled implantable pulse generators (e.g., Medtronic Percept™) and undergo standardized DBS programming assessments. The intervention of interest includes DBS parameter testing combined with recording of local field potentials (LFPs) and patient-reported subjective ratings using a visual analogue scale (VAS). Clinical assessments and neuroimaging data are integrated to identify personalized stimulation "sweet spots" and to evaluate the relationship between subjective symptom improvement and electrophysiological biomarkers.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — No intervention (observational study)

SUMMARY:
This multicenter, prospective and retrospective diagnostic study investigates personalized programming strategies for deep brain stimulation (DBS) in patients with Parkinson's disease. DBS of the subthalamic nucleus (STN) is an established therapy for advanced Parkinson's disease; however, optimization of stimulation parameters remains time-consuming and resource-intensive due to the growing complexity of electrode designs and programming options.

The PERCEPT-DBS study aims to improve DBS programming by combining subjective patient-reported outcomes with objective electrophysiological biomarkers. Specifically, the study examines the relationship between patients' subjective assessment of stimulation efficacy, measured using a visual analogue scale (VAS), and local field potentials (LFPs), with a focus on beta-band activity recorded from implanted DBS electrodes. These data are integrated with structural and functional neuroimaging to identify individualized stimulation "sweet spots" within the STN.

A total of 24 patients with idiopathic Parkinson's disease treated with bilateral STN-DBS will be recruited across several German DBS centers. Participants undergo standardized clinical assessments, VAS-based blinded monopolar reviews, and LFP recordings using sensing-enabled implantable pulse generators. In addition, imaging-based analyses are performed to relate electrophysiological and subjective measures to anatomical and connectomic features.

The primary objective is to determine whether electrophysiological markers correlate with subjective patient ratings and whether their overlap defines personalized optimal stimulation targets. By integrating patient perception with neurophysiological and imaging data, this study seeks to advance individualized DBS programming strategies and contribute to the development of more efficient, patient-centered, and potentially adaptive DBS therapies.

ELIGIBILITY:
Inclusion Criteria:

Age between 35 and 80 years

Clinically confirmed idiopathic Parkinson's disease according to Movement Disorder Society (MDS) criteria

Status post bilateral deep brain stimulation of the subthalamic nucleus (STN-DBS)

Implanted DBS system suitable for electrophysiological recordings (prospective cohort: sensing-enabled IPG)

Ability to understand study procedures and communicate reliably with the investigator

Written informed consent provided

Exclusion Criteria:

Any condition impairing the ability to provide informed consent or comply with study procedures

Presence of exclusion criteria for Parkinson's disease according to MDS criteria

Manifest dementia according to ICD-10 criteria

Severe neurological, psychiatric, or medical conditions interfering with study participation or assessments

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients with idiopathic Parkinson's disease treated with bilateral subthalamic nucleus deep brain stimulation (STN-DBS). Participants are recruited from specialized DBS centers during postoperative follow-up or ambulatory care. All patients are capable of providing informed consent and participating in standardized clinical, electrophysiological, and patient-reported assessments. The cohort includes individuals implanted with DBS systems that allow recording of local field potentials, enabling analysis of electrophysiological biomarkers in relation to subjective patient-reported DBS efficacy and neuroimaging data.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between beta-band local field potentials and patient-reported DBS efficacy | 30 to 45 days after DBS electrode implantation (first study visit)
  The primary outcome is the relationship between electrophysiological activity recorded from the subthalamic nucleus and subjective patient assessment of deep brain stimulation (DBS) efficacy. Beta-band (13-30 Hz) local field potential (LFP) amplitude recorded from implanted DBS electrodes is correlated with patient-reported ratings of overall stimulation quality measured using a visual analogue scale (VAS) during blinded monopolar programming. Outcome analyses assess whether electrophysiological markers correspond to higher subjective DBS benefit and whether overlapping signals define individualized stimulation "sweet spots."

CONTACTS AND LOCATIONS:
Locations (1):
- LMU University Hospital, München, Germany

IPD SHARING:
Plan to Share IPD: No